CLINICAL TRIAL: NCT01987401
Title: CSP #595Pilot - Respiratory Health and Deployment to Iraq and Afghanistan Pilot
Brief Title: Service and Health During the Iraq and Afghanistan Era
Acronym: CSP #595 Pilot
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 595Pilot
Record Dates: First submitted 2013-11-12; First posted 2013-11-19 (Estimated); Results first posted 2018-09-12 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Iraq and Afghanistan Era Veterans
Keywords: pulmonary; lung; military and environmental exposures; epidemiologic; observational; interview or questionnaire; deployment related; Enduring Freedom; Iraqi Freedom

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 50 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Iraq and Afghanistan Era Veterans: Veterans who served during the Iraq and Afghanistan Era

SUMMARY:
The primary objective of CSP #595, "Service and Health During the Iraq and Afghanistan Era," is to characterize the impact of deployment to Iraq and Afghanistan on the respiratory health of Veterans. The purpose of the pilot study is to determine the willingness of Veterans who served during the Iraq and Afghanistan Era to provide health and military service information. This information will help us design a larger national study.

DETAILED DESCRIPTION:
The primary objective of CSP #595, "Respiratory Health and Deployment to Iraq and Afghanistan," is to assess the association of airborne exposures encountered during deployment with current measures of respiratory health among U.S. military Veterans who served in Iraq and Afghanistan.

The purpose of the pilot study is to assess the feasibility and approach to conducting a large, multi-site Cooperative Studies Program (CSP) initiative to characterize the impact of deployment to Iraq and Afghanistan on the respiratory health of Veterans. The investigators will (a) determine the most efficient and feasible method for recruitment; (b) understand demographic, health-related, and military service-related factors influencing participation so that potential biases can be identified; and (c) demonstrate that the proposed individual exposure reconstruction techniques based on deployment history are feasible.

Three aims are proposed: Aim 1: Using the Department of Defense (DoD) Defense Manpower Data Center (DMDC) master personnel roster, identify a representative sample of deployed Veterans who have served in Iraq and Afghanistan as well as a sample of non-deployed Veterans; identify the optimal methods for recruitment of participants to Phase 1 of data collection (mailed survey or telephone interview on self-reported health and military service history) and assess the willingness of Veterans to visit a nearby Veterans Health Administration (VHA) medical center to participate in Phase 2 in-person data collection, which includes more extensive self-reported health information, lifetime exposure ascertainment, and assessment of pulmonary function. Aim 2: Assess the Phase 2 participation rate of Veterans using VA Boston Healthcare System as a pilot study site. Aim 3: Using publically available exposure data and data from the DoD personnel file, demonstrate that the proposed individual exposure reconstruction techniques are feasible.

The study is organized by the CSP Epidemiology Center program with the Seattle Epidemiologic Research and Information Center serving as the CSP coordinating center. The 2 participating sites are at the VA Boston Healthcare System and Durham VA Medical Center. The pilot study will provide information that will allow the planning of a national, large-scale health study to assess the residual effects of exposure to high levels of particulate matter while deployed. This will help inform VA health policy for Iraq and Afghanistan Veterans.

ELIGIBILITY:
Inclusion Criteria:

* All competent, living men and women who served during the Iraq and Afghanistan Era and been discharged from the Army, Air Force, Marine Corps, or Navy are eligible to participate.
* Individuals in respective Guard and Reserve units are also eligible to participate.
* A Veteran is eligible without regard to deployment or combat status and without regard to current or past user status in the Veterans Health Administration.

Exclusion Criteria:

* Veterans of the Coast Guard, including individuals in respective Guard and Reserve units, are not eligible to participate.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Veterans who served during the Iraq and Afghanistan Era, without regard to actual deployment, identified from the Department of Defense (DoD) Defense Manpower Data Center (DMDC) master personnel roster of all persons serving during the time period of interest.
Sampling Method: Probability Sample
Enrollment: 1242 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Garshick, MD, Study Chair — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA; Rebecca B McNeil, PhD, Study Chair — Durham VA Medical Center, Durham, NC; Susan P Proctor, DSc, Study Chair — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (2):
- United States (2):
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Click here for more information about this study: CSP #595Pilot - Respiratory Health and Deployment to Iraq and Afghanistan Pilot — http://www.seattle.eric.research.va.gov/
- See also: Click here for more information about this study: CSP #595Pilot - Respiratory Health and Deployment to Iraq and Afghanistan Pilot — http://www.research.va.gov/programs/csp/

RESULTS

PARTICIPANT FLOW:
Groups:
- Mailed Survey: Participants who received the survey by mail.
- Telephone Survey: Participants who received the survey by telephone.
- In-person Survey: Participants who received survey in person.
Period: Overall Study
Arm/Group | Mailed Survey | Telephone Survey | In-person Survey
Started | 591 | 591 | 60
Completed | 137 | 121 | 16
Not Completed | 454 | 470 | 44

BASELINE CHARACTERISTICS:
Groups:
- Mail: Received mail survey
- Phone: Received phone survey
- In-Person: Invited to in-person survey
- Total: Total of all reporting groups
Arm/Group | Mail | Phone | In-Person | Total
Number analyzed (Participants) | 591 | 591 | 60 | 1242
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (10.9) | 39.4 (11.5) | 36.7 (10.6) | 38.7 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 93 | 8 | 188
  Male | 504 | 498 | 52 | 1054
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 5 | 0 | 10
  Asian | 24 | 22 | 3 | 49
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 89 | 97 | 3 | 189
  White | 452 | 449 | 51 | 952
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 21 | 18 | 3 | 42
Region of Enrollment [Number; unit: participants]
  United States | 591 | 591 | 60 | 1242

OUTCOME MEASURES:

1. Primary Outcome: Participation Rates
Description: From the national sample, the investigators will compare participation rates for the mailed survey and telephone survey. Among a sample of Veterans living in the greater Boston area, the investigators will calculate participation rate for the in-person survey.
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mailed Survey | Telephone Survey | In-person Survey
Number analyzed (Participants) | 591 | 591 | 60
Participants | 137 | 121 | 14

ADVERSE EVENTS:
Arm/Group | Mailed Survey | Telephone Survey | In-person Survey
All-Cause Mortality (participants affected / at risk) | 0/591 | 0/591 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/591 | 0/591 | 0/60
Other Adverse Events (participants affected / at risk) | 0/591 | 0/591 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No